CLINICAL TRIAL: NCT05632588
Title: Near Fatal Asthma in Children and Young People
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC22026
Record Dates: First submitted 2022-10-25; First posted 2022-11-30 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Near Fatal Asthma
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational surveillance study

SUMMARY:
This study will report the frequency, risks factors, clinical care and estimate the future asthma risk of children and young people (aged 5-15 years) experiencing a Delphi defined near fatal asthma (NFA) attacks in the United Kingdom (UK) and Republic of Ireland (ROI). A greater understanding of the frequency and risk factors associated with NFA could help support children and young people (CYP), parents and clinicians to identify and modify risk, both independently and through a resulting clinical care pathway and also develop future research to improve effectiveness of interventions. The study will explore both commonly identified clinical factors, but also for the first time describe in detail the variance in medical management (acute and intensive care) that could lead to future clinical trials and guideline development to standardise care. The study will also describe, through data-linkage, socio-demographic factors associated with NFA, to include pollution, pollen, weather, viral prevalence that could lead to better care for higher risk CYP.

To encourage more consistent, less fragmented care following a near fatal asthma attack, the study will consider how care is provided subsequent to an NFA attack using British Paediatric Surveillance Unit (BPSU) surveillance at 12 and 24 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* A child/young person is considered to have experienced an episode of near fatal asthma if they meeting any one of the following:

  1. Any child aged 5-15 years surviving* an acute episode of asthma, who when presenting self-ventilating with severe dyspnoea (e.g. inability to speak) and all the following features:

     1. Pulse oxygen saturation below 92% despite maximal oxygen therapy (i.e. 10-15l/min oxygen flow via non-rebreather mask) during acute presentation
     2. pH <= 7.2 and/or pCO2 >=60mmHg or 8kPa
     3. Escalation to use of intravenous bronchodilator infusion
  2. Any child aged 5-15 years surviving* an acute episode of asthma, who had a respiratory arrest and/or required cardiopulmonary resuscitation as part of their presentation.
  3. Any child age 5-15 years surviving* an acute episode of asthma for which he/she was invasively ventilated.

     * surviving to hospital discharge

Exclusion Criteria:

* CYP not meeting the case definition will be excluded. An expert panel (consisting of three clinicians) will adjudicate borderline cases.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The number of children and young people identified who experience NFA within the 18-month surveillance period is not known, but is estimated to be c400 (from paediatric intensive care admission data). All UK and ROI hospitals where children may attend with acute asthma could be potential contributing sites. Each case will be followed up for 24 months following the near fatal asthma event.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of cases of Near Fatal Asthma reported to British Paediatric Surveillance Unit | 18 months
  Descriptive data

SECONDARY OUTCOMES:
Detailed analysis of the clinical, social and environmental characteristics of those who experience NFA. | 18 months
  Descriptive data
Detailed analysis of the care provided to CYP who experience NFA at the time of the event, during emergency, in patient and critical care. | 18 months
  Descriptive data
Reporting of the 12 and 24 months following an episode of NFA, estimating the future risk of a health-related asthma event and the healthcare that is provided to those experiencing NFA. | 42 months
  Descriptive data

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No